CLINICAL TRIAL: NCT06585540
Title: A Pilot Study to Evaluate Barhemsys for the Prevention of Postoperative Nausea and Vomiting in the Bariatric Surgery Population
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Principal Investigator, Justin Liberman, Staff Anesthesiologist, Department of Anesthesia, Benaroya Research Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CRP23057
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Post Operative Nausea and Vomiting
Keywords: Post Operative Nausea and Vomiting; Bariatric Surgery; Bariatric; Barhemsys; Amisulpride
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, subject blinded, placebo-controlled crossover pilot study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group Barhemsys (Experimental): Interventional arm receiving Barhemsys during surgery
  Interventions: Drug: Amisulpride IV Prevention
- Group Placebo (Placebo Comparator): Placebo arm receiving Placebo during surgery
  Interventions: Drug: Placebo Preventative
- Group Placebo Barhemsys (Experimental): Of patients who are members of Group Placebo they will be able to receive Barhemsys in the Post Anesthesia Care Unit if they experience nausea or emesis
  Interventions: Drug: Amisulpride IV Treatment
- Group Placebo Placebo (Placebo Comparator): Of patients who are members of Group Placebo they will be able to receive Placebo in the Post Anesthesia Care Unit if they experience nausea or emesis
  Interventions: Drug: Placebo Treatment

INTERVENTIONS:
Drug: Amisulpride IV Prevention — Patients in this arm will receive Amisulpride 5mg IV as a preventative dose after the induction of anesthesia
  Other Names: Amisulpride IV Treatment
  Arms: Group Barhemsys
Drug: Amisulpride IV Treatment — Patients in this arm will receive Amisulpride 10mg IV for first-line treatment of Post-Operative Nausea and Vomiting in the post-anesthesia care unit.
  Arms: Group Placebo Barhemsys
Drug: Placebo Preventative — Patients in this arm will receive placebo (Normal Saline) while under general anesthesia
  Arms: Group Placebo
Drug: Placebo Treatment — Patients in this Arm will receive placebo as first line treatment of Post-Operative Nausea and Vomiting in the Post Anesthesia Care Unit
  Arms: Group Placebo Placebo

SUMMARY:
To assess the effectiveness of Amisulpride to treat Post Operative Nausea and Vomiting (PONV) and to assess the effectiveness of Amisulpride to prevent PONV following bariatric surgery.

DETAILED DESCRIPTION:
This is a phase III/IV, randomized, placebo-controlled, patient-blinded cross-over pilot study to evaluate the effectiveness of Amisulpride in the treatment and prevention of Post Operative Nausea and Vomiting (PONV) in adult patients, 18-65 years of age, at a single surgery site in the pacific northwest who are undergoing bariatric surgery. Approximately 100 patients will be randomized in a 1:1 ratio to receive a single intravenous dose of Amisulpride (5mg IV single dose) or a placebo (saline control, 1mL IV single dose) at the induction of anesthesia. Those who initially receive placebo will undergo an additional randomization in the post-anesthesia care unit (PACU) to receive a dose of Amisulpride (10mg IV single dose) or placebo (saline control, 2mL IV single dose) in a 1:1 ratio as first line treatment for PONV.

ELIGIBILITY:
Inclusion Criteria:

* The study will recruit adult patients (Age 18-65) scheduled for bariatric surgery. Additional inclusion criteria include ASA class I-III and patients who plan to be inpatient for at least 24 hours.

Included Surgeries:

Robotic, Laparoscopic or Open Roux-en-Y Robotic, Laparoscopic or Open Gastric Sleeve Robotic, Laparoscopic or Open Gastrectomy Robotic, Laparoscopic or Open Revision Gastric Bypass

Exclusion Criteria:

* Pregnant or breastfeeding
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Congenital QTc abnormalities
* Current use of droperidol
* Parkinson's disease
* Allergy to Barhemsys
* GFR < 30 mL/min/1.73m2
* Emergency surgery or add-on cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With "Complete Response" in the Post Anesthesia Care Unit | Until Patient Leaves Post Anesthesia Care Unit (60-120 minutes)
  Complete response is defined as no occurrence of vomiting or retching, no nausea score ≥ 1 and no use of rescue medication during their Post Anesthesia Care Unit stay.

SECONDARY OUTCOMES:
Incidence of complete response to established Post-operative Nausea and Vomiting | Until Patient leave Post Anesthesia Care Unit (60-90 minutes)
  Effectiveness of Barhemsys in the treatment of established nausea or vomiting in the high-risk bariatric surgical population during Post Anesthesia Care Unit stay. Failure of complete response is defined as subject emesis or use of rescue medication during Post Anesthesia Care Unit stay following a treatment dose of Barhemsys.
Number of participants with no nausea | Up to 24 hours following surgery
  Nausea (defined as the desire to vomit without the presence of expulsive muscular movements) measured on a 0-10 verbal response scale, where 0=no nausea at all and 10=the worst nausea imaginable. "No nausea" means no score ≥ 1.
Number of Participants with no Emesis | Up to 24 hours following surgery
  Emesis is defined as vomiting (production of even the smallest amount of stomach contents) or retching (muscular movements of vomiting but without expulsion of stomach contents, usually because of an empty stomach)
Number of Participants With no Use of Rescue Medication | Up to 24 hours following surgery
  Any agent given in the post-operative period with the intention of providing anti-emetic rescue is counted as rescue antiemetic medication for the purposes of efficacy determination, even if it did not achieve control of emesis or was given incorrectly (e.g., wrong dosage or route). Any agent given in the postoperative period which would be expected, by virtue of its pharmacology, dosage, and route, to exert a clinically meaningful antiemetic effect was considered as rescue antiemetic medication, even if administered inadvertently or without the intention of providing rescue.
The Number of Participants With no Emesis, no Significant Nausea, and no Use of Rescue Medication | Up to 24 hours following surgery
  No occurrence of vomiting/retching, no nausea score ≥ 4 on verbal response scale (where 0=no nausea at all and 10=the worst nausea imaginable) and no use of rescue medication.
The Number of Participants With no Significant Nausea | Up to 24 hours following surgery
  Nausea (defined as the desire to vomit without the presence of expulsive muscular movements) measured on a 0-10 verbal response scale, where 0=no nausea at all and 10=the worst nausea imaginable. "No significant nausea" means no score ≥ 4.

CONTACTS AND LOCATIONS:
Overall Officials: Justin S Liberman, Medical Doctor, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share IPD would only be required if the researches felt that information could be used to improve patient safety. This information would be shared with the FDA.

REFERENCES:
- [Background] Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010 Feb;104(2):158-66. doi: 10.1093/bja/aep370. Epub 2009 Dec 26. PMID 20037151
- [Background] Berger ER, Huffman KM, Fraker T, Petrick AT, Brethauer SA, Hall BL, Ko CY, Morton JM. Prevalence and Risk Factors for Bariatric Surgery Readmissions: Findings From 130,007 Admissions in the Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program. Ann Surg. 2018 Jan;267(1):122-131. doi: 10.1097/SLA.0000000000002079. PMID 27849660
- [Background] Habib AS, Kranke P, Bergese SD, Chung F, Ayad S, Siddiqui N, Motsch J, Leiman DG, Melson TI, Diemunsch P, Fox GM, Candiotti KA. Amisulpride for the Rescue Treatment of Postoperative Nausea or Vomiting in Patients Failing Prophylaxis: A Randomized, Placebo-controlled Phase III Trial. Anesthesiology. 2019 Feb;130(2):203-212. doi: 10.1097/ALN.0000000000002509. PMID 30475232
- [Background] Candiotti KA, Kranke P, Bergese SD, Melson TI, Motsch J, Siddiqui N, Chung F, Rodriguez Y, Minkowitz HS, Ayad SS, Diemunsch P, Fox G. Randomized, Double-Blind, Placebo-Controlled Study of Intravenous Amisulpride as Treatment of Established Postoperative Nausea and Vomiting in Patients Who Have Had No Prior Prophylaxis. Anesth Analg. 2019 Jun;128(6):1098-1105. doi: 10.1213/ANE.0000000000003733. PMID 31094774
- [Background] Fox GM, Albayaty M, Walker JL, Xue H, Darpo B. Intravenous Amisulpride Does Not Meaningfully Prolong the QTc Interval at Doses Effective for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2021 Jan;132(1):150-159. doi: 10.1213/ANE.0000000000004538. PMID 31913911
- [Background] Apfel CC, Philip BK, Cakmakkaya OS, Shilling A, Shi YY, Leslie JB, Allard M, Turan A, Windle P, Odom-Forren J, Hooper VD, Radke OC, Ruiz J, Kovac A. Who is at risk for postdischarge nausea and vomiting after ambulatory surgery? Anesthesiology. 2012 Sep;117(3):475-86. doi: 10.1097/ALN.0b013e318267ef31. PMID 22846680
- [Background] Carroll NV, Miederhoff P, Cox FM, Hirsch JD. Postoperative nausea and vomiting after discharge from outpatient surgery centers. Anesth Analg. 1995 May;80(5):903-9. doi: 10.1097/00000539-199505000-00009. PMID 7726432
- [Background] White PF, O'Hara JF, Roberson CR, Wender RH, Candiotti KA; POST-OP Study Group. The impact of current antiemetic practices on patient outcomes: a prospective study on high-risk patients. Anesth Analg. 2008 Aug;107(2):452-8. doi: 10.1213/ane.0b013e31817b842c. PMID 18633023
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- See also: FDA label for Amisulpride — https://www.accessdata.fda.gov/drugsatfda_docs/label/2020/209510s000lbl.pdf